CLINICAL TRIAL: NCT00392873
Title: "REFUEL" Active Women's Study II: Increased Caloric Intake to Reverse Energy Deficiency in Exercising Women: Impact on Bone and Menstrual Cyclicity
Brief Title: Increased Calorie Intake to Reverse Energy Deficiency in Exercising Women: Impact on Bone and Menstrual Cyclicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary Jane DeSouza, Professor of Kinesiology and Physiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15353
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Menstrual Irregularity
Keywords: Amenorrhea; Energy deficiency; Resting energy expenditure; Bone metabolism; Bone mineral density; Exercise
MeSH Terms: conditions — Menstruation Disturbances; Amenorrhea; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EAMD+Calories (Experimental): This group contains women with exercise-associated menstrual disturbances (EAMD) and receives an intervention of increased caloric intake during the 12-month intervention. The targeted increase in caloric intake is 20-30% of baseline energy expenditure.
  Interventions: Behavioral: EAMD+Calories
- EAMD Control (No Intervention): This group contains women with exercise-associated menstrual disturbances (EAMD) and undergoes the same procedures as the EAMD+Calories group. However, this group is instructed to maintain exercise and eating habits.
- Heathy Control (No Intervention): This group contains exercising women with regular, ovulatory menstrual cycles. this group is instructed to maintain body weight and exercise and eating habits.

INTERVENTIONS:
Behavioral: EAMD+Calories — During the 12 month intervention, volunteers in the Increased calorie intake group will follow a modified dietary plan designed to achieve and maintain a target level of 20-30% above their previously determined baseline, in an effort to achieve a chronic energy surplus of +20-30% over their baseline energy requirements.
  Arms: EAMD+Calories

SUMMARY:
The purpose of this study is to examine the effects of increased food intake on the menstrual cycle and bone health in physically active women who have irregular or absent menstrual cycles. This study will examine whether a 12 month period of increased food intake will cause menstrual cycles to resume and help bones get stronger.

DETAILED DESCRIPTION:
Low levels of estrogen found in physically active, premenopausal women with irregular or absent menstrual periods is likely caused by insufficient energy (calorie) intake compared to energy expenditure. Premenopausal women with menstrual disturbances and amenorrhea suffer from reductions in bone mineral density, particularly in the lumbar spine. Bone loss observed in amenorrheic women may be serious enough to result in osteoporotic fractures, but is also associated with a high prevalence of stress fractures. Increased calorie intake should help improve energy status, menstrual status, and bone health.

Comparison: Premenopausal women with irregular or absent menstrual periods will be assigned to either receive additional calories or serve as controls. A group of premenopausal women with normal menstrual periods will also be used for comparison.

ELIGIBILITY:
Inclusion Criteria for Ovulatory Control Volunteers:

* 18-35 years
* BMI 16-25 kg/m2
* At least 2 hr/wk of aerobic exercise
* Gynecological age >/= 5 years
* Weight stable (+/- 2 kg) last 6 months
* History of regular menses for 6 months

Inclusion Criteria for Women with Irregular or Absent Menses:

* 18-35 years
* BMI 16-25 kg/m2
* At least 3 hr/wk of aerobic exercise
* Gynecological age >/= 5 years
* Weight stable (+/- 2 kg) last 6 months
* No menses within past 3 months or 6 or less menses in last 12 months
* Low to normal bone mass (L1-L4 Z score </=0)

Exclusion Criteria for all participants:

* Hormonal contraceptives in last 6 months
* Smoking currently
* Current clinical diagnosis of an eating disorder
* Use of medications incompatible with measurement of reproductive or metabolic hormones, including thyroid medications that may interfere with any of the study outcomes.
* Dietary habits incompatible with prescribed diet for study
* Any metabolic, reproductive or bone disease
* Sedentary individuals with less than 120 minutes (2 hrs) of activity per week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 233 (Actual)
Dates: Start 2006-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reproductive hormones | 1 year
Metabolic hormones | 1 year
Metabolic bone markers | 1 year
Bone mineral density | 1 year

SECONDARY OUTCOMES:
Eating Disorder Inventory-2 (EDI-2) | 1 year
Three Factor Eating Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane De Souza, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Women's Health and Exercise Laboratories, The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Strock NCA, De Souza MJ, Mallinson RJ, Olmsted M, Allaway HCM, O'Donnell E, Plessow F, Williams NI. 12-months of increased dietary intake does not exacerbate disordered eating-related attitudes, stress, or depressive symptoms in women with exercise-associated menstrual disturbances: The REFUEL randomized controlled trial. Psychoneuroendocrinology. 2023 Jun;152:106079. doi: 10.1016/j.psyneuen.2023.106079. Epub 2023 Mar 8. PMID 36947969
- [Derived] De Souza MJ, Ricker EA, Mallinson RJ, Allaway HCM, Koltun KJ, Strock NCA, Gibbs JC, Kuruppumullage Don P, Williams NI. Bone mineral density in response to increased energy intake in exercising women with oligomenorrhea/amenorrhea: the REFUEL randomized controlled trial. Am J Clin Nutr. 2022 Jun 7;115(6):1457-1472. doi: 10.1093/ajcn/nqac044. PMID 35170727
- [Derived] De Souza MJ, Mallinson RJ, Strock NCA, Koltun KJ, Olmsted MP, Ricker EA, Scheid JL, Allaway HC, Mallinson DJ, Kuruppumullage Don P, Williams NI. Randomised controlled trial of the effects of increased energy intake on menstrual recovery in exercising women with menstrual disturbances: the 'REFUEL' study. Hum Reprod. 2021 Jul 19;36(8):2285-2297. doi: 10.1093/humrep/deab149. PMID 34164675
- [Derived] Southmayd EA, Williams NI, Mallinson RJ, De Souza MJ. Energy Deficiency Suppresses Bone Turnover in Exercising Women With Menstrual Disturbances. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3131-3145. doi: 10.1210/jc.2019-00089. PMID 30896746